CLINICAL TRIAL: NCT06393270
Title: 5-year Clinical Follow-up of Bulk-fill Restorative Materials in Class II Restorations
Brief Title: 5-year Clinical Follow-up of Restorative Materials
Status: Completed | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Merve Gurses, Assistant Professor, Selcuk University
Other Study IDs: SelcukD
Record Dates: First submitted 2024-04-24; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Dental Caries; Class II Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Equia Forte Fil: High-viscosity glass ionomer cement
  Interventions: Diagnostic Test: Modified US Public Health Service (USPHS) criteria
- Tetric Bulk Fill: Bulk-fill composite material
  Interventions: Diagnostic Test: Modified US Public Health Service (USPHS) criteria
- Filtek Bulk Fill: Bulk-fill composite material
  Interventions: Diagnostic Test: Modified US Public Health Service (USPHS) criteria

INTERVENTIONS:
Diagnostic Test: Modified US Public Health Service (USPHS) criteria — Dental caries classification system

SUMMARY:
Materials to be used as permanent filling materials in Class II restorations are still an essential field of study. This study aims to evaluate the 5-year clinical performance of Class II restorations performed with different bulk-fill restorative materials.

The study was planned as an observational clinical trial. In the study, Class II restorations performed with Tetric Bulk Fill (TBF) and Filtek Bulk Fill (FBF) composites and Equia Forte Fil (EF) will be evaluated. Fifty-one patients and 119 restorations will be included in the study. Restorations will be assessed in terms of modified United States Public Health Service (USPHS) criteria during the 5th year. Cochran Q, Pearson chi-square, and Fisher-Freeman-Halton tests will be used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were;

  1. older than 18 years old
  2. had good general health and oral hygiene
  3. had interface restorations of similar size in their premolars and molars
  4. were able to attend control appointments were included The teeth were determined as follows;

  <!-- -->

  1. in contact with the opposing tooth
  2. exposed to normal occlusal forces on the dentition
  3. restoration width not exceeding 1⁄2 of the intercuspal distance
  4. normal response to vitality tests without periodontal pathology

Exclusion Criteria:

* Patients with;

  1. poor oral hygiene
  2. those with active periodontal disease
  3. those with severe bruxism
  4. pregnant and lactating women
  5. endodontically treated teeth were excluded from the study

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: Seventy-nine patients (50 females, 29 males) between the ages of 18 and 53, and 192 restorations meeting the criteria were included in the study.
Sampling Method: Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Retention | 5th year.
  At the control appointment, it was determined whether there was material loss in the restoration. The scale used includes the characters A, B, and C. A is the best clinical result.
Color Match | 5th year.
  At the control appointment, it was determined whether the restoration's color harmony with the adjacent tooth tissue was maintained. The scale used includes the characters A, B, and C. A is the best clinical result.
Marginal Adaptation | 5th year.
  At the follow-up appointment, it was determined whether there was any deterioration in the marginal adaptation of the restoration. The scale used includes the characters A, B, and C. A is the best clinical result.
Marginal Discoloration | 5th year.
  At the control appointment, it was determined whether there was any color change at the edges of the restoration. The scale used includes the characters A, B, and C. A is the best clinical result.
Secondary Caries | 5th year.
  At the follow-up appointment, it was determined whether there was any decay under the restoration. The scale used includes the characters A and C. A is the best clinical result.
Surface Texture | 5th year.
  At the control appointment, it was determined whether the restoration surface had a defect. The scale used includes the characters A, B, and C. A is the best clinical result.
Anatomical Form | 5th year.
  At the control appointment, it was determined whether the restoration maintained its anatomical form. The scale used includes the characters A, B, and C. A is the best clinical result.
Postoperative Sensitivity | 5th year.
  At the follow-up appointment, it was determined whether there was postoperative sensitivity after the restorative procedure. The scale used includes the characters A, B, and C. A is the best clinical result.

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Faculty of Dentistry, Konya, Turkey (Türkiye)

REFERENCES:
- [Derived] Gurses M, Inan B, Cobanoglu N, Turkmen ATK. Five-year clinical follow-up of bulk-fill restorative materials in class II restorations. Dent Mater J. 2024 Sep 28;43(5):746-754. doi: 10.4012/dmj.2024-132. Epub 2024 Sep 10. PMID 39261021